CLINICAL TRIAL: NCT07307820
Title: Sutureless Glueless Technique Versus Interrupted Suturing for Conjunctival Autograft Fixation After Primary Pterygium Excision: Anterior Segment Optical Coherence Tomography (ASOCT) Study
Acronym: ASOCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mahmoud Ramadan, lecturer of ophthalmolgy, Minia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 166072025
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Primary Pterygium, ASOCT, Conjunctival Autograft Surgery
Keywords: Primary pterygium, ASOCT, conjunctival autograft surgery

STUDY DESIGN:
Intervention Model Description: Randomized contralateral-eye design, where each patient contributed both eyes, one receiving sutured and the other sutureless graft fixation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sutured conjunctival autograft fixation (Experimental): conjunctival autograft secured with interrupted 10/0 nylon after pterygium exision
  Interventions: Procedure: sutured conjunctival autograft fixation
- sutureless glueless conjunctival autograftfixation (Experimental): Conjunctival autograft placed without sutures, relying on natural adhesion and fibrin clot formation.
  Interventions: Procedure: Sutureless Conjunctival Autograft Fixation

INTERVENTIONS:
Procedure: sutured conjunctival autograft fixation — After pterygium excision, a conjunctival autograft is secured in place using interrupted 10-0 nylon sutures to ensure graft stability and promote healing
  Arms: sutured conjunctival autograft fixation
Procedure: Sutureless Conjunctival Autograft Fixation — Following pterygium excision, the conjunctival autograft is placed without sutures, relying on natural adhesion and fibrin clot formation to maintain graft position.
  Arms: sutureless glueless conjunctival autograftfixation

SUMMARY:
This study aims to compare the clinical and Anterior segment optical coherence tomography (ASOCT) outcomes between sutured and sutureless conjunctival autograft fixation techniques in the management of primary pterygium.

A total of 30 patients with bilateral primary pterygia were included. Each patient underwent pterygium excision in both eyes: one eye received graft fixation using interrupted 10-0 nylon sutures, while the fellow eye received sutureless fixation. Allocation of technique between eyes was randomized.

All surgeries were performed by the same surgeon, and patients were followed up weekly for one month. Parameters assessed included graft thickness, interface reflectivity, gutter size, conjunctival congestion, donor site healing, and postoperative discomfort using a visual analogue scale.

The study evaluates which fixation method provides faster healing, better cosmetic results, and fewer complications such as graft slippage or recession, especially in relation to pterygium size.

ELIGIBILITY:
Inclusion Criteria Age 18 to 65 years (both sexes). Diagnosis of bilateral primary nasal pterygium requiring surgical excision (both eyes affected).

Horizontal corneal encroachment of the pterygium ≥ 2.0 mm in each eye. Lesions amenable to conjunctival autograft coverage with expected graft size obtainable from superior bulbar conjunctiva.

Willingness and ability to attend scheduled follow-up visits for 1 month postoperatively.

Able to provide written informed consent.

Exclusion Criteria Recurrent pterygium in either eye. Previous ocular surgery on the study eye(s) (including prior pterygium surgery) or conjunctival grafting.

Active ocular surface disease or infection (e.g., conjunctivitis, keratitis) at screening.

Severe dry eye disease (e.g., Schirmer's test ≤ 5 mm or TBUT < 5 s) likely to affect healing.

Significant ocular comorbidities affecting wound healing or outcome interpretation: uncontrolled glaucoma with conjunctival filtering surgery, ocular surface cicatrizing disorders (e.g., ocular pemphigoid), severe blepharitis, or severe meibomian gland dysfunction.

Systemic conditions that impair wound healing or increase surgical risk (e.g., uncontrolled diabetes mellitus with HbA1c > 8.0%, connective tissue disorders, immunosuppression, chronic systemic corticosteroid use).

Current use of anticoagulant therapy that cannot be safely paused per local perioperative protocol (if this precludes safe graft fixation).

Pregnancy or breastfeeding. Known allergy to any material used in the procedure or postoperative medications.

Inability to comply with follow-up schedule or provide informed consent (e.g., cognitive impairment, planning to move away).

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Graft stability: incidence of slippage or recession (%) - Secondary (Safety/Complication) | Time Frame: Within 1 month postoperatively
  Proportion of eyes with clinically significant graft slippage or marginal recession requiring intervention or observed during follow-up.
Patient-reported discomfort (VAS 0-10) - Secondary | Time Frame: Day 1, Week 1, Week 2, Week 3, Week 4
  Mean Visual Analogue Scale (0 = no discomfort to 10 = worst possible) recorded at each visit.
Cosmetic outcome - surgeon-rated score (0-10) | Time Frame: 4 weeks (Month 1) postoperatively
  Surgeon's cosmetic grading based on redness, graft contour and surface smoothness (0 = poor to 10 = excellent).

SECONDARY OUTCOMES:
Interface reflectivity (qualitative grading: low/moderate/high) | Time Frame: Week 1, Week 2, Week 3, Week 4
  Qualitative grading of graft-host interface reflectivity on AS-OCT to indicate edema/fibrosis; images assessed by masked grader(s).
Change in central graft thickness (µm) - | Baseline (Day 1) to Week 4
  Absolute and percent change in central graft thickness from Day 1 to Week 4 measured by AS-OCT.
Mean central graft thickness measured by AS-OCT (µm) | Time Frame: 4 weeks (Month 1) postoperatively
  Description: Mean central conjunctival autograft thickness measured by anterior-segment OCT at 4 weeks after surgery. Measurement performed using device calipers on the central graft area; reported as mean ± SD per group. This endpoint assesses final early structural integration and resolution of postoperative edema.
Conjunctival congestion score (0-3) | Time Frame: Day 1, Week 1, Week 2, Week 3, Week 4
  Clinician-graded vascular hyperemia (0 = none; 1 = mild; 2 = moderate; 3 = severe) at each visit.
Gutter size at graft-host junction (µm) | Time Frame: Week 1, Week 2, Week 3, Week 4
  Linear measurement of the graft-host interface gap (gutter) by AS-OCT at each follow-up; reported as mean ± SD.
Operative time (minutes) - Secondary | Time Frame: At surgery (intraoperative)
  Duration from incision to completion of graft fixation, recorded in minutes for each eye.
Early recurrence (clinical evidence of fibrovascular regrowth at limbus) - | Time Frame: 4 weeks (Month 1) postoperatively
  Presence or absence of early fibrovascular regrowth onto cornea at 1 month (noting that longer follow-up is required for definitive recurrence rates).
Adverse events (type and severity) - Secondary (Safety) | Time Frame: Within 1 month postoperatively
  All adverse events related to the procedure recorded and graded (e.g., infection, granuloma, graft loss), with details on management
Donor site epithelialization (complete: Y/N and time to healing in days) - Secondary | Time Frame: Assessed weekly up to 4 weeks
  Presence of complete re-epithelialization of donor site confirmed clinically and by AS-OCT; record time (days) to complete healing.

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University Hospital, Minya, Minia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to institutional policies regarding patient privacy and confidentiality, as well as restrictions based on ethical committee requirements. Data sharing may be reconsidered upon formal request and in compliance with all relevant regulations protecting participant information."

REFERENCES:
- [Background] Natung T, et al. Sutureless, glue-less conjunctival autograft versus sutured autograft in primary pterygium surgery. PMC article. 2017
- [Background] Mahajan S, et al. A Comparative Study of Suture-less and Glue-Free versus Sutured Conjunctival Autograft in Pterygium Surgery. Arch of Medical & Health Science. 2021
- [Background] Aguilar-Gonzalez M, Espana-Gregori E, Pascual-Camps I, Gomez-Lechon-Quiros L, Peris-Martinez C. Prospective Study: Utility of Anterior Segment Optical Coherence Tomography to Identify Predictive Factors of Recurrence in Pterygium Surgery. J Clin Med. 2024 Aug 14;13(16):4769. doi: 10.3390/jcm13164769. PMID 39200911